CLINICAL TRIAL: NCT01073358
Title: Resection of Colorectal Liver Metastases With or Without Routine Hilar Lymphadenectomy - A Randomized Controlled Trial
Brief Title: Resection of Colorectal Liver Metastases With or Without Routine Hilar Lymphadenectomy
Acronym: RELY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Nuh Rahbari, PD MD, University Hospital Carl Gustav Carus
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NNR-5
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Hepatic Metastases; Colorectal Cancer
Keywords: resectable hepatic metastases of colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: No routine hilar lymphadenectomy (No Intervention): Resection of colorectal liver metastases without routine hilar lymphadenectomy
- Group B: Routine hilar lymphadenectomy (Experimental): Hilar lymphadenectomy is performed before actual resection of the colorectal liver metastases.
  Interventions: Procedure: Routine hilar lymphadenectomy

INTERVENTIONS:
Procedure: Routine hilar lymphadenectomy — Hilar lymphadenectomy is performed before actual resection of the colorectal liver metastases
  Arms: Group B: Routine hilar lymphadenectomy

SUMMARY:
It is uncertain, whether hilar lymphadenectomy should be performed routinely in patients undergoing resection of colorectal liver metastases.

For this reason it is the aim of the present prospective randomized trial to evaluate, if routine lymphadenectomy reduces recurrent disease in patients undergoing resection of colorectal liver metastases.

DETAILED DESCRIPTION:
Routine lymphadenectomy in patients undergoing hepatic resection for colorectal liver metastases may improve outcome of further patients due to the presence of micrometastases that have been shown to be of prognostic relevance. While previous studies highlight the clinical significance of perihepatic lymph node metastases, the outcome of patients with and without hilar lymphadenectomy has not yet been compared and thus no clear conclusion about the clinical value of routine hilar lymphadenectomy in CRC patients undergoing resection of liver metastases can be drawn from present data.

As disease recurrence occurs frequently and may affect up to 75 % of patients, further strategies are required to improve postoperative outcome. Routine hilar lymphadenectomy may offer an effective approach to remove residual disease and by this to reduce disease recurrence with little additional morbidity. For this reason it is the aim of the present prospective randomized trial to evaluate, if routine lymphadenectomy reduces recurrent disease in patients undergoing resection of colorectal liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for curative (R0) resection
* No evidence of extrahepatic disease
* No history of previous hepatic lymphadenectomy
* Age equal or greater than 18 years
* Written Informed consent

Exclusion Criteria:

* Expected lack of compliance
* Impaired mental state or language problems
* History of another primary cancer, except:

  * Curatively treated in situ cervical cancer or curatively resected non-melanoma skin cancer
  * Other primary solid tumour curatively treated with no known active disease present and no treatment administered for ≥ 5 years prior to randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2010-03-09 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
rate of disease recurrence | 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Weitz, MD, MSc, Principal Investigator — Department of Gastrointestinal, Thoracic and Vascular Surgery Dresden
Locations (1):
- Department of Gastrointestinal, Thoracic and Vascular Surgery, Dresden, Germany